CLINICAL TRIAL: NCT03574064
Title: Investigation of GLP-2 Mechanism of Action
Brief Title: Effects of Gut Peptides on Bone Remodeling
Acronym: KS-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirsa Skov-Jeppesen, Principal Investigator, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UCPH-KS-3-18
Record Dates: First submitted 2018-06-07; First posted 2018-06-29 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — Incretins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GLP-2 (Experimental): Glucagon-Like Peptide-2 (GLP-2)
  Interventions: Other: Glucagon-Like Peptide-2 (GLP-2)
- GIP (Experimental): Glucose-dependent Insulinotropic polypeptide (GIP)
  Interventions: Other: Glucose-dependent insulinotropic polypeptide (GIP)
- GLP-2+GIP (Experimental): GLP-2+GIP
  Interventions: Other: GLP-2+GIP
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Glucagon-Like Peptide-2 (GLP-2) — Glucagon-Like Peptide-2 (GLP-2) injection.
  Arms: GLP-2
Other: Glucose-dependent insulinotropic polypeptide (GIP) — Glucose-dependent insulinotropic polypeptide (GIP) injection.
  Arms: GIP
Other: GLP-2+GIP — GLP-2+GIP injection.
  Arms: GLP-2+GIP
Other: Placebo — Placebo injection.
  Arms: Placebo

SUMMARY:
We will investigate effects of gut hormones on bone remodeling.

ELIGIBILITY:
Inclusion Criteria:

Women Age above 50 years Postmenopausal Caucasian BMI 18.5 to 28.0 kg/m2.

Exclusion Criteria:

Smoking Medication believed to influence study outcome Weight change more than 3 kg whitin the last 3 months Overweight surgery Intestinal surgery Hgb<7,0 mmol/L Decreased renal function

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
C-terminal telopeptide (CTX). At all time points and AUC(0-240 min). | -10 minutes to 600 minutes
  CTX is a marker of bone resorption. Measured in serum.
N-terminal propeptide of type 1 procollagen (P1NP). At all time points and AUC(0-240 min). | -10 minutes to 600 minutes
  P1NP is a marker of bone formation. Measured in serum.

SECONDARY OUTCOMES:
PTH | -10 minutes to 600 minutes
  Bone marker. Measured in serum.
Sclerostin | -10 minutes to 600 minutes
  Bone marker.
Calcium | -10 minutes to 600 minutes
  Measured in serum within 5 days.
Glucose | -10 minutes to 600 minutes
  Measured in serum.
Glucose-dependent insulinotropic polypeptide (GIP) | -10 minutes to 600 minutes
  Total and intact GIP. Measured in plasma.
Insulin | -10 minutes to 600 minutes
  Measured in serum.
C-peptide | -10 minutes to 600 minutes
  Measured in serum.
Glukagon-like peptide-1 (GLP-1) | -10 minutes to 600 minutes
  Measured in plasma.
Glucagon | -10 minutes to 600 minutes
  Measured in plasma.
Glukagon-like peptide-2 (GLP-2) | -10 minutes to 600 minutes
  Intact GLP-2. Measured in plasma.
PP | -10 minutes to 600 minutes
  Measured in plasma.

OTHER OUTCOMES:
Blood pressure | -10 minutes to 60 minutes
  Measured before blood sampling.
Heart rate | -10 minutes to 60 minutes
  Measured before blood sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided